CLINICAL TRIAL: NCT01942538
Title: Study of the Effectiveness of Maintenance rTMS Sessions for 6 Months Versus Placebo in Subjects With Fibromyalgia Responders to 3 Week-rTMS Treatment
Brief Title: Efficiency of Repetitive Transcranial Magnetic Stimulation (rTMS) Sessions After a Successful 3 Week-treatment in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Jean-Christophe Dumont, Medical Doctor, Assistant in Rheumatologia Service CHU Limoges, Centre Hospitalier Esquirol
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013-A00820-45
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Fibromyalgia
Keywords: rTMS; fibromyalgia; sham; maintenance session; pain
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- rTMS-rTMS (Experimental): subjects receiving real rTMS treatment and real rTMS maintenance sessions
  Interventions: Device: rTMS
- sham - sham (Sham Comparator): subjects receiving sham treatment and presenting a clinical improvement : they will be submitted to sham maintenance sessions
  Interventions: Device: sham rTMS
- rTMS-sham (Sham Comparator): subjects receiving sham rTMS maintenance sessions after successful real rTMS treatment
  Interventions: Device: rTMS; Device: sham rTMS
- rTMS (Experimental): real rTMS for 3 weeks but without clinical improvement
  Interventions: Device: rTMS
- sham (Sham Comparator): sham treatment for 3 weeks without clinical improvement
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: rTMS — one session : 20 runs of 10 seconds high frequency stimulation(10Hz) and 50 seconds pause - power equivalent to 90% of the motor threshold
  Arms: rTMS; rTMS-rTMS; rTMS-sham
Device: sham rTMS — same session as defined with the real rTMS, but with a coil not delivering magnetic field.
  Arms: rTMS-sham; sham; sham - sham

SUMMARY:
Maintenance rTMS sessions after a successful 3week-rTMS treatment for subjects with fibromyalgia may maintain the clinical improvement.

DETAILED DESCRIPTION:
In a previous pilot study, a 3 week treatment with rTMS in fibromyalgia subjects induced a 40% improvement of pain feeling. Three months later, the pain level was still significantly reduced in comparison with the beginning of the treatment, but the clinical improvement was less than at the end of the treatment. We thus propose to realize real or sham rTMS sessions at 3 weeks interval during 6 months with subjects presenting a significant clinical improvement after a 3 week-rTMS or sham treatment to evaluate the response maintenance.

ELIGIBILITY:
Inclusion Criteria:

* presence of the criteria from the American College of Rheumatology (2010)for fibromyalgia diagnosis,
* painful state for more than six months,
* visual analogic scale evaluation > or = 5,
* age between 18 and 70,
* no modification in therapeutic treatment one month before and during the protocol
* presence of actual or prior antalgic chronic treatment : pregabalin, duloxetine, milnacipran, gabapentin, venlafaxine, laroxyl, grade 1 or 2 antalgic
* residence in Limoges or the periphery, or the ability to come to the hospital for the treatment

Exclusion Criteria:

* presence of non stabilized psychiatric comorbidity (personality trouble, addiction, suicide attempt, non controlled affective trouble),
* active epilepsy,
* previous cerebral traumatism, or cerebral surgery, intra-cranial hyper tension,
* pacemaker, metallic pieces in the brain, cochlear ocular implant, or any metallic material contra indicating magnetic resonance imaging.
* clozapine, bupropion, methadon, theophyllin, or other non chemical antalgic technic established during the previous month(kinesitherapy, relaxation, hypnosis...),
* pregnancy, or administrative and judiciary protection, absence of health insurance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-09; Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
number of fibromyalgia subjects maintaining a clinical improvement with rTMS maintenance sessions during 6 months | 210 days
  = number of fibromyalgia subjects maintaining a clinical improvement after a prior rTMS treatment (15 sessions in 3 weeks)and maintenance rTMS sessions administered at 42, 63, 84, 105, 126, 147, 168, 189, 210 days after inclusion in comparison with sham maintenance sessions.
  clinical improvement is described as a 30% decrease from baseline in pain feeling (visual analogue scale) and a response ≥ 6 for the Patient's global impression of Change.
  effect will be considered as maintained if criteria of clinical improvement present after 3 week rTMS treatment are conserved at 6 months rTMS or sham maintenance sessions.

SECONDARY OUTCOMES:
number of rTMS responders at 3week-rTMS treatment | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Dumont, MD, Principal Investigator — CHU Dupuytren CH Esquirol
Locations (2):
- France (2):
  - Centre Hospitalier Esquirol, Limoges
  - Centre Hospitalier Universitaire, Limoges

REFERENCES:
- [Background] Ciobanu C, Girard M, Marin B, Labrunie A, Malauzat D. rTMS for pharmacoresistant major depression in the clinical setting of a psychiatric hospital: effectiveness and effects of age. J Affect Disord. 2013 Sep 5;150(2):677-81. doi: 10.1016/j.jad.2013.03.024. Epub 2013 May 11. PMID 23673085